CLINICAL TRIAL: NCT01210547
Title: Assessment of Dental, Skeletal Pattern, and Soft Tissue Using Three-dimensional Images
Brief Title: Three-dimensional Assessment of Craniofacial Structures
Status: Terminated | Type: Observational
Why Stopped: Lack of funding, departure of key personnel
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 0912M75577
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this project is to reduce the radiation exposure in orthodontic patients by the use of a new imaging protocols based on non-ionizing orthodontic records (e.g. digital dental models, three-dimensional photograph) The first step in this process is to develop and validate an orthodontic analysis able to assess craniofacial proportions, dental, skeletal, and facial soft tissue. The investigators working hypothesis is that data from three-dimensional facial photographs and from digital dental casts can be registered accurately and consistently, and the diagnostic information about tooth position and facial soft-tissue derived from them are comparable to x-ray derived data

ELIGIBILITY:
Inclusion Criteria:

* Full permanent dentition
* Complete set of digital orthodontic records
* Must be able to follow directions

Exclusion Criteria:

* Incomplete orthodontic records

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Current patients attending the University of Minnesota School of Dentistry Orthodontic Clinic, and who voluntarily agreed to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2010-09; Primary Completion 2013-10 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Assessment of dental and soft tissue position relative to cone-beam computed tomography (CBCT) | At the time of initial orthodontic records

CONTACTS AND LOCATIONS:
Overall Officials: Brent E Larson, DDS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Orthodontic Clinic, Minneapolis, Minnesota, United States